CLINICAL TRIAL: NCT04749810
Title: Prospective Observational Study of Long-term Pathogenic Treatment of Elizaria® in Patients With Atypical Hemolytic Uremic Syndrome
Brief Title: Observational Study of Elizaria® in aHUS Patients
Status: Completed | Type: Observational
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Other Study IDs: ECU-aHUS-N01
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-02

CONDITIONS: Atypical Hemolytic Uremic Syndrome; aHUS
Keywords: Atypical Hemolytic Uremic Syndrome; Azotemia; Hemolytic-Uremic Syndrome; Hemolysis; Syndrome; Disease; Pathologic Processes; Uremia; Kidney Diseases; Urologic Diseases; Anemia, Hemolytic; Anemia; Hematologic Diseases; Thrombotic Microangiopathies; Thrombocytopenia; Blood Platelet Disorders
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome; Azotemia; Hemolytic-Uremic Syndrome; Hemolysis; Syndrome; Disease; Pathologic Processes; Uremia; Kidney Diseases; Urologic Diseases; Anemia, Hemolytic; Anemia; Hematologic Diseases; Thrombotic Microangiopathies; Thrombocytopenia; Blood Platelet Disorders | interventions — eculizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elizaria®: Eculizumab
  Interventions: Drug: Elizaria®

INTERVENTIONS:
Drug: Elizaria® — Induction cycle: 900 mg (3 vials of 30 mL, 10 mg/mL) intravenous infusion for 30 minutes once a week for 4 weeks. Maintenance therapy: 1200 mg (4 vials of 30 mL, 10 mg/mL) intravenous infusion for 30 minutes in Week 5, followed by 1200 mg every 14 days.
  Other Names: Eculizumab

SUMMARY:
It is a multicenter observational non-comparative study of the efficacy and safety of long-term pathogenetic Elizaria® therapy in patients with atypical Hemolytic Uremic Syndrome

DETAILED DESCRIPTION:
After screening, patients meeting all of the inclusion / non-inclusion criteria and vaccinated against meningococcal infections were treated by Elizaria®.

The study is planned to include at least 50 patients receiving Elizaria® for the aHUS treatment.

The study will consist of a screening period of up to 4 weeks, including, if necessary, immunization with meningococcal vaccine, a treatment period of 52 weeks.

Medication will be prescribed in accordance with routine medical practice. Accordingly to minimize the risks and subjectivity of assessments the methods adopted in the routine practice of treating patients with aHUS will be used.

Investigators enroll patients with aHUS diagnosis who have indications for pathogenetic therapy and who are receiving Elizaria® under the government program. Patients will receive medication in accordance with the established requirements of national standards and protocols for the treatment of patients with aHUS. The registration of the amount of the drug used will be carried out on the basis of information in the Patient Diaries, as well as primary documentation.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent to study participation.
2. Male and female patients aged 2 months and older with documented atypical hemolytic uremic syndrome (aHUS)diagnosis.
3. By the time of inclusion in the study, Elizaria® should be prescribed as a pathogenetic therapy for aHUS; Exclusion Criteria

1. Intolerance to eculizumab, or other components of the drug.

Min Age: 2 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: At least 50 adult and pediatric patients (from 2 months), with a confirmed diagnosis of aHUS, who meet the enrollment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in platelet count compared to the screening level | 52 week
  Change in platelet count at 52 week after treatment with study drug compared to baseline at screening

SECONDARY OUTCOMES:
Change in lactate dehydrogenase (LDH) levels from baseline at screening | 52 week
  Change in LDH levels at 52 week after starting study drug treatment from baseline at screening
Proportion of patients with normalized platelet levels | 52 week
  Proportion of patients with normal platelet count at 52 week after initiation of study drug treatment
Proportion of patients with no thrombotic microangiopathy (TMA) events | 52 week
  The absence of TMA-related events is defined as the absence, for at least 12 weeks, of: 1) a decrease in platelet counts greater than 25% from baseline at screening; 2) plasma therapy; 3) hemodialysis.
Proportion of TMA-related interventions | 52 week
  The proportion of TMA-related interventions is defined as (number of plasma therapy sessions + number of hemodialysis sessions) / number of patient days.
Proportion of patients with complete TMA response | 52 week
  Complete TMA response is defined as the absence of abnormalities in LDH and platelet levels + improvement in renal function (decrease in creatinine levels by 25% or more compared to the baseline value on screening) when performed at least two consecutive tests within 8 weeks
Change in eGFR (ml / min. / 1.73m2) compared with the baseline level at screening; | 52 week
  Change in eGFR (mL/min/1.73m2) at 52 week after initiation of study drug treatment from baseline at screening
Proportion of patients with an improvement in glomerular filtration rate (eGFR) of 15 ml / min / 1.73m2 or more compared to the baseline level at screening. | 52 week
  Proportion of patients with improvement in eGFR of 15 ml/min/1.73m2 or more at 52 week after treatment with study drug compared to baseline at screening
Proportion of patients with more then 1 stage-improvement in chronic kidney desease (CKD) compared to baseline at screening. | 52 week
  Proportion of patients with >=1 stage improvement in CKD at 52 week after initiation of study drug treatment compared with baseline at screening
Proportion of patients with an increase in hemoglobin level of more than 20 g / l compared to the baseline level at screening. | 52 week
  Proportion of patients with an increase in hemoglobin level of more than 20 g/l at 52 week after the start of study drug treatment compared with baseline at screening
Dynamics of membrane attack complex (MAC) level compared to baseline at Visit 2 | 52 week
  Changes in MAC levels at 52 week compared to baseline
The frequency and severity of adverse events (AEs) | 52 weeks
  Frequency and severity of adverse events (AEs), including serious adverse events (SAEs) and AEs associated with study drug use
Proportion of patients with antidrug antibodies | 52 weeks
  Proportion of patients with antidrug antibodies; titer of antidrug antibodies and their neutralizing activity

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — AO GENERIUM
Locations (8):
- Russia (8):
  - Federal State Budgetary Educational Institution of Higher Education "Kazan State Medical University" of the Ministry of Health of the Russian Federation, Kazan'
  - Regional State Budgetary Healthcare Institution "Krasnoyarsk' Regional Clinical Center for Maternity and Childhood Protection", Krasnoyarsk
  - State budgetary healthcare institution of the city of Moscow "Children's City Clinical Hospital of St. Vladimir of the Healthcare Department of the City of Moscow", Moscow
  - Federal State Autonomous Educational Institution of Higher Education "First Moscow State Medical University n.a. I.M. Sechenov" of the Ministry of Health of the Russian Federation, Moscow
  - State budgetary healthcare institution of the City of Moscow "City clinical hospital #52 of the Moscow City Healthcare Department", Moscow
  - State budgetary healthcare institution of the city of Moscow "City Clinical Hospital n.a. A.K. Eramishantsev of the Moscow City Healthcare Department", Moscow
  - St. Petersburg's State Budgetary Healthcare Institution "City Mariinsky Hospital", Saint Petersburg
  - St. Petersburg's State Budgetary Healthcare Institution "Children's City Multidisciplinary Clinical Specialized Center of High Medical Technologies", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No